CLINICAL TRIAL: NCT06292663
Title: Can Preoperative Information Via Virtual Reality Affect Patient's Anxiety? A Randomized Controlled Trial and Patient Interviews
Brief Title: Can Preoperative Information Via Virtual Reality Affect Patient's Anxiety?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EMN-2023-08767
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Surgery; Pain
Keywords: Virtual Reality; VR; Distraction; Non-pharmacological; Total Knee Arthroplasty; Orthopedic surgery; Orthopaedics; Spinal Anesthesia; Readiness
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The subjects are being randomized to one of two groups.
Who Masked: Investigator
Masking Description: The primary investigator will stay blinded in this study and an assistant to the investigator is screening and including the patients and collecting data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients allocated to this group are getting the standard information from their anesthesiologist and a supplement of information via. a Virtual Reality (VR) headset. The information they get through the VR headset is about their course on the day of their surgery.
  Interventions: Device: Virtual Reality
- Control Group (No Intervention): Patients allocated to this group are only getting standard information from their anesthesiologist.

INTERVENTIONS:
Device: Virtual Reality — The subjects get a supplement of information via. a Vitual Reality (VR) headset. The information they get through the VR headset is about their course on the day of their surgery.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to test and learn about Virtual Reality (VR) providing preoperative information to patients undergoing elective TKA surgery in spinal anesthesia. The main question(s) aim(s) to answer if:

* Can preoperative information through a VR headset lower the patients preoperative anxiety?
* Can VR information make the patients more ready for surgery. Painscore will also be collected.

Participants will be randomized into two groups. One that will have preoperative information through VR versus standard information.

If there is a comparison group: Researchers will compare enrolled TKA patients to see if VR have an impact on anxiety, readiness and pain

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) causes pain, disability and poor quality of life in the elderly. Consequently, it can severely affect people's quality of life and physical function. International guidelines recommend exercise therapy alongside patient education and weight management (if needed) as first-line treatment for all individuals with knee OA. However, more than 1,000,000 TKA procedures are performed annually worldwide, and with aging populations and an increase in obesity, this number is expected to increase markedly4. Although TKA is generally considered an effective treatment option, up to 20% of patients are not fully satisfied after surgery5. Spinal anesthesia is commonly used during primary TKA given the purported safety benefits, quicker immediate postoperative recovery, decreased intraoperative bleeding, and lower transfusion rates when compared to general anesthesia. To help the patient feel more comfortable and relaxed during a procedure, administration of sedative medication titrated by the anesthetist is common practice. Despite a low rate of complications associated with spinal anesthesia compared to general anesthesia, it is important to acknowledge that complications can still occur.

Virtual Reality (VR) demonstrates signs as a promising tool to support healthcare, including mentally preparing the patient for a surgical procedure. Preoperative readiness, expectations, anxiety, and pain perception are crucial to the patient's surgical experiences. VR can immerse patients into a virtual environment and distract patients from e.g., unpleasant sounds, sights, and feelings. Integrating VR into preoperative care has shown the potential to offer several advantages, such as promoting patients' distraction, knowledge, and information. However, harms have been reported such as cyber sickness but only in few cases among older adult patients.

Offering a controlled environment where patients can familiarize themselves with the surgical process through VR shown on a head-mounted display (HMD) and with sound reduction headphones provides them an opportunity to explore, e.g., the operation theater, waiting area, and PACU.

All this can foster a sense of confidence and increased readiness and lead to an overall improved patient experience.

Ethical considerations: this trial will assess the effects of using a VR patient journey preoperatively. Therefore, the trial will be highly systematic and at low risk of producing biased results. The trial will be adequately powered to limit the risk of random error. The participants receiving standard of care will likely not benefit directly from the trial. However, the participants in the control group will potentially assist with valuable evidence, which might benefit future patients. Participants can, at any time, for any reason, withdraw their consent to participate in the trial. If participants withdraw from the trial, it will not impact the level of care and treatment offered by the departments.

Informed consent: the trial will be conducted according to national and international standards of Good Clinical Practice. This trial protocol and amendments will be submitted to the Committee on Health Research Ethics in the Region Zealand of Denmark for approval before initiation of the trial. All patients scheduled for total knee arthroplasty will be screened for inclusion. The patients will be provided oral and written information about the trial, including potential benefits and risks, and invited to participate. The oral and written information will enable the patient to decide whether or not to participate in the trial. If the patients match all inclusion criteria and none of the exclusion criteria and decides to participate in the trial, both the patient and one of the trial personnel will have to sign the written informed consent paper.

The oral and written information can be provided by the Ph.D. student, a project nurse, or any employee from the project, collectively known as "trial personnel." The trial personnel can obtain consent. The trial personnel will be trained in all the procedures related to screening, informing potential participants, obtaining informed consent and inclusion of participants, randomization of participants, and how to handle the VR equipment.

Patients scheduled for elective surgery will be informed about the conduct of the trial at the anesthesia or orthopedic pre-consult, and written trial information will be provided.

All patients considered for inclusion will be informed about the mandatory verbal trial information consult. The patients will be informed of the possibility of bringing a next of kin to the mandatory verbal trial information consult. The verbal trial information consult will be held by other personnel trained to do so according to the Good Clinical Practice guidelines. The consult will take place in an explicit reserved room to prevent any disruptions. . The patient will be informed of the possibility of considering participation in the trial. The verbal trial information consult will be based on written information and contain information on the trial's purpose, potential risks and benefits, and the conduct of the trial. We will ensure that all patients, irrespective of being scheduled for surgery, will have at least 24 hours to consider their participation in the trial.

The patient will be informed that participation in the trial is voluntary and that consent can be withdrawn at any time without the decision to withdraw impacting further treatment. The patient will be asked if the investigators may continue to collect data relevant to the trial from the patient's medical records and if we are allowed to call them postoperatively to schedule an interview. Patients will be informed that randomization takes place on the day when the pre-anesthetic meeting is taking place. All stakeholders are bound by secrecy. The patient will receive trial information and the written informed consent declaration.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for total knee arthroplasty
* Scheduled for spinal anesthesia
* Age of 18 or above
* Ability to understand the trial protocol, risks, and benefits and provide signed informed consent

Exclusion Criteria:

* Inability to read and understand Danish
* Uncooperativeness (as judged by investigators)
* Claustrophobia or fear of small spaces
* Disorders that prevent the person from wearing a VR device
* Highly visually or auditive impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | On the 1 day of inclusion and on the 1 day of the patient's surgery
  Anxiety will be measured by using The Amsterdam Preoperative Anxiety and Information Scale (APAIS). The questionnaire contains six questions addressing topics: worries about the anesthetic, need for information about the anesthetic, worries about the procedure, and need for information about the procedure. Furthermore, the patients fill out the Numerical Rating Scale (NRS) according to anxiety rating from 0-10. 0 is no anxiety at alle, and 10 is the worst imaginable anxiety.

SECONDARY OUTCOMES:
Cumulative sedative consumption | On the 1 day of the patient's surgery
  Cumulative sedation is the total amount of sedatives administrated before and during surgery, and all sedative medications will be collected for comparison. Different opioids will be converted to morphine IV equivalents for comparison. The information will be collected from the digital patient journal (Sundhedsplatformen) by one of the research assistant.
Opioid consumption | On the 1 day of the patient's surgery
  We will assess opioid consumption by conducting data from the digital patient journal (Sundhedsplatformen).
Patient preoperatively expectations | On the 1 day of inclusion
  The Treatment Expectation Questionnaire (TEX-Q) will assess patient expectation preoperatively. The questionnaire contains 15 questions and six supplemental questions dealing with; expected benefits, expected positive and negative impact, expected harm, desired benefits, desired impact, feared harm, feared negative impact, process-related expectations, and expected behavioral control of the treatment.
Patient preoperatively readiness | On the 1 day of inclusion and on the 1 day of the patient's surgery
  Readiness will be measured using the Preoperative Assessment of Readiness Tool (PART). The questionnaire contains 15 questions about readiness: understanding consent to the operation, time to ask questions, understanding the benefit of surgery, staff confirmation, enough time to decide, social security, spiritual preparation, and economic preparation.
Adverse events | From the beginning of the intervention and until the end of the intervention period (48 hours postoperatively).
  Adverse events are defined as any unwanted event, sign, or symptom occurring during the trial, whether the adverse is related to the VR head-mounted display or not. All adverse events will be noted in the Case Report Form. Adverse events are considered related to the trial from randomization until the end of the intervention period (48 hours postoperatively). The assumed adverse event's beginning, end, severity, and symptoms will be noted.

OTHER OUTCOMES:
Level of pain | On the 1 day of inclusion and the 1 day of the patient's surgery, at PACU and 24 hour postoperatively
  Pain will be assessed at the day of inclusion, at the day of surgery, at the Post Anesthesia Care Unit (PACU), and 24hr after surgery (+/- 4hr). The research assistant will ask the patient to rate their pain on a scale from 0-10. 0 is no pain, and 10 is the worst imaginable pain.
The need for information | On the 1 day of inclusion and on the 1 day of the patient's surgery
  The need for information among patients will be assesed by using the The Amsterdam Preoperative Anxiety and Information Scale (APAIS)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Geisler, phd, Study Director — Region Hovedstadens Apotek
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. BMC Musculoskelet Disord. 2017 Feb 7;18(1):72. doi: 10.1186/s12891-017-1439-y. PMID 28173795
- [Background] Rupp M, Lau E, Kurtz SM, Alt V. Projections of Primary TKA and THA in Germany From 2016 Through 2040. Clin Orthop Relat Res. 2020 Jul;478(7):1622-1633. doi: 10.1097/CORR.0000000000001214. PMID 32168057
- [Background] Dunbar MJ, Richardson G, Robertsson O. I can't get no satisfaction after my total knee replacement: rhymes and reasons. Bone Joint J. 2013 Nov;95-B(11 Suppl A):148-52. doi: 10.1302/0301-620X.95B11.32767. PMID 24187375
- [Background] Lu Y, Cregar WM, Goodloe JB, Khazi Z, Forsythe B, Gerlinger TL. General Anesthesia Leads to Increased Adverse Events Compared With Spinal Anesthesia in Patients Undergoing Unicompartmental Knee Arthroplasty. J Arthroplasty. 2020 Aug;35(8):2002-2008. doi: 10.1016/j.arth.2020.03.012. Epub 2020 Mar 12. PMID 32247674
- [Background] Hoxhallari E, Behr IJ, Bradshaw JS, Morkos MS, Haan PS, Schaefer MC, Clarkson JHW. Virtual Reality Improves the Patient Experience during Wide-Awake Local Anesthesia No Tourniquet Hand Surgery: A Single-Blind, Randomized, Prospective Study. Plast Reconstr Surg. 2019 Aug;144(2):408-414. doi: 10.1097/PRS.0000000000005831. PMID 31348351
- [Background] Torres GCS, Fernandez DF, Ledbetter L, Relf MV. Systematic Review of Preoperative Patient Readiness. AORN J. 2021 Jul;114(1):47-59. doi: 10.1002/aorn.13425. PMID 34181266
- [Background] Chang SL, Kuo MJ, Lin YJ, Chen SA, Chen CT, Yang YY, Yang LY, Kao SY, Shulruf B, Lee FY. Virtual reality-based preprocedural education increases preparedness and satisfaction of patients about the catheter ablation of atrial fibrillation. J Chin Med Assoc. 2021 Jul 1;84(7):690-697. doi: 10.1097/JCMA.0000000000000555. PMID 34029219
- [Background] Drazich BF, McPherson R, Gorman EF, Chan T, Teleb J, Galik E, Resnick B. In too deep? A systematic literature review of fully-immersive virtual reality and cybersickness among older adults. J Am Geriatr Soc. 2023 Dec;71(12):3906-3915. doi: 10.1111/jgs.18553. Epub 2023 Aug 10. PMID 37560978
- [Background] Tharion JG, Kale S. Patient Satisfaction Through an Immersive Experience Using a Mobile Phone-Based Head-Mounted Display During Arthroscopic Knee Surgery Under Spinal Anesthesia: A Randomized Clinical Trial. Anesth Analg. 2021 Oct 1;133(4):940-948. doi: 10.1213/ANE.0000000000005666. PMID 34283040
- [Background] Vaughn F, Wichowski H, Bosworth G. Does preoperative anxiety level predict postoperative pain? AORN J. 2007 Mar;85(3):589-604. doi: 10.1016/S0001-2092(07)60130-6. PMID 17352896
- [Background] Wilson JM, Farley KX, Erens GA, Guild GN 3rd. General vs Spinal Anesthesia for Revision Total Knee Arthroplasty: Do Complication Rates Differ? J Arthroplasty. 2019 Jul;34(7):1417-1422. doi: 10.1016/j.arth.2019.03.048. Epub 2019 Mar 28. PMID 31005435
- [Background] Eberhart L, Aust H, Schuster M, Sturm T, Gehling M, Euteneuer F, Rusch D. Preoperative anxiety in adults - a cross-sectional study on specific fears and risk factors. BMC Psychiatry. 2020 Mar 30;20(1):140. doi: 10.1186/s12888-020-02552-w. PMID 32228525
- [Background] Zemla AJ, Nowicka-Sauer K, Jarmoszewicz K, Wera K, Batkiewicz S, Pietrzykowska M. Measures of preoperative anxiety. Anaesthesiol Intensive Ther. 2019;51(1):64-69. doi: 10.5603/AIT.2019.0013. PMID 31280554
- [Background] Clarke IM, Barnes D. Depression and anxiety in pain clinics. Anaesthesia. 1986 Mar;41(3):325-6. doi: 10.1111/j.1365-2044.1986.tb12802.x. No abstract available. PMID 3963341
- [Background] Walker EMK, Bell M, Cook TM, Grocott MPW, Moonesinghe SR; Central SNAP-1 Organisation; National Study Groups. Patient reported outcome of adult perioperative anaesthesia in the United Kingdom: a cross-sectional observational study. Br J Anaesth. 2016 Jun 12;117(6):758-766. doi: 10.1093/bja/aew381. PMID 27956674
- [Background] Wang R, Huang X, Wang Y, Akbari M. Non-pharmacologic Approaches in Preoperative Anxiety, a Comprehensive Review. Front Public Health. 2022 Apr 11;10:854673. doi: 10.3389/fpubh.2022.854673. eCollection 2022. PMID 35480569
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Bhugaonkar K, Bhugaonkar R, Masne N. The Trend of Metaverse and Augmented & Virtual Reality Extending to the Healthcare System. Cureus. 2022 Sep 12;14(9):e29071. doi: 10.7759/cureus.29071. eCollection 2022 Sep. PMID 36258985
- [Background] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] Chuan A, Zhou JJ, Hou RM, Stevens CJ, Bogdanovych A. Virtual reality for acute and chronic pain management in adult patients: a narrative review. Anaesthesia. 2021 May;76(5):695-704. doi: 10.1111/anae.15202. Epub 2020 Jul 27. PMID 32720308
- [Background] Felemban OM, Alshamrani RM, Aljeddawi DH, Bagher SM. Effect of virtual reality distraction on pain and anxiety during infiltration anesthesia in pediatric patients: a randomized clinical trial. BMC Oral Health. 2021 Jun 25;21(1):321. doi: 10.1186/s12903-021-01678-x. PMID 34172032
- [Background] Lier EJ, Oosterman JM, Assmann R, de Vries M, van Goor H. The effect of Virtual Reality on evoked potentials following painful electrical stimuli and subjective pain. Sci Rep. 2020 Jun 3;10(1):9067. doi: 10.1038/s41598-020-66035-4. PMID 32494060
- [Background] Chan Z, Kan C, Lee P, Chan I, Lam J. A systematic review of qualitative studies: patients' experiences of preoperative communication. J Clin Nurs. 2012 Mar;21(5-6):812-24. doi: 10.1111/j.1365-2702.2011.03942.x. Epub 2011 Oct 18. PMID 22008151
- [Background] Tipotsch-Maca SM, Varsits RM, Ginzel C, Vecsei-Marlovits PV. Effect of a multimedia-assisted informed consent procedure on the information gain, satisfaction, and anxiety of cataract surgery patients. J Cataract Refract Surg. 2016 Jan;42(1):110-6. doi: 10.1016/j.jcrs.2015.08.019. PMID 26948785
- [Background] Shukla AN, Daly MK, Legutko P. Informed consent for cataract surgery: patient understanding of verbal, written, and videotaped information. J Cataract Refract Surg. 2012 Jan;38(1):80-4. doi: 10.1016/j.jcrs.2011.07.030. Epub 2011 Nov 6. PMID 22062774
- [Background] Fakes KL, Hall AE, Carey ML, Boyes AW, Symonds M, Evans TJ, Sanson-Fisher RW. Development and Validation of the MiPrep Survey: An Instrument Assessing Patients' Perceived Preparation for Medical Interventions Including Medical Imaging, Radiotherapy, and Surgery. Value Health. 2019 Jun;22(6):704-711. doi: 10.1016/j.jval.2019.01.017. Epub 2019 May 17. PMID 31198188
- [Background] Torres GCS, Relf MV, Tuazon JA. The mediating role of pre-operative patient readiness on surgical outcomes: A structural equation model analysis. J Adv Nurs. 2020 Jun;76(6):1371-1383. doi: 10.1111/jan.14339. Epub 2020 Mar 18. PMID 32128862
- [Background] Torres GCS, Macindo JRB. Scale Development and Psychometric Evaluation of the Preoperative Assessment of Readiness Tool. J Perianesth Nurs. 2018 Dec;33(6):895-907. doi: 10.1016/j.jopan.2016.07.010. PMID 30449438
- [Background] Conner-Spady BL, Marshall DA, Hawker GA, Bohm E, Dunbar MJ, Frank C, Noseworthy TW. You'll know when you're ready: a qualitative study exploring how patients decide when the time is right for joint replacement surgery. BMC Health Serv Res. 2014 Oct 2;14:454. doi: 10.1186/1472-6963-14-454. PMID 25278186
- [Background] Phillips AW, Horgan AF. Fast track surgery and preoperative optimization. Surg (United Kingdom) 2014; 32: 84-8.
- [Background] Rajabiyazdi F, Alam R, Pal A, Montanez J, Law S, Pecorelli N, Watanabe Y, Chiavegato LD, Falconi M, Hirano S, Mayo NE, Lee L, Feldman LS, Fiore JF Jr. Understanding the Meaning of Recovery to Patients Undergoing Abdominal Surgery. JAMA Surg. 2021 Aug 1;156(8):758-765. doi: 10.1001/jamasurg.2021.1557. PMID 33978692
- [Background] Gunaratne R, Pratt DN, Banda J, Fick DP, Khan RJK, Robertson BW. Patient Dissatisfaction Following Total Knee Arthroplasty: A Systematic Review of the Literature. J Arthroplasty. 2017 Dec;32(12):3854-3860. doi: 10.1016/j.arth.2017.07.021. Epub 2017 Jul 21. PMID 28844632
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035
- [Background] Hawker GA, Conner-Spady BL, Bohm E, Dunbar MJ, Jones CA, Ravi B, Noseworthy T, Dick D, Powell J, Paul P, Marshall DA; BEST-Knee Study Team. Patients' Preoperative Expectations of Total Knee Arthroplasty and Satisfaction With Outcomes at One Year: A Prospective Cohort Study. Arthritis Rheumatol. 2021 Feb;73(2):223-231. doi: 10.1002/art.41510. Epub 2020 Dec 26. PMID 32892511
- [Background] Jones CA, Suarez-Almazor ME. Patient expectations and total knee arthroplasty. J Clin Outcomes Manag 2017; 24: 364-70.
- [Background] Frisaldi E, Shaibani A, Benedetti F. Why We should Assess Patients' Expectations in Clinical Trials. Pain Ther. 2017 Jun;6(1):107-110. doi: 10.1007/s40122-017-0071-8. Epub 2017 May 5. PMID 28477082
- [Background] Mira JJ, Tomas O, Virtudes-Perez M, Nebot C, Rodriguez-Marin J. Predictors of patient satisfaction in surgery. Surgery. 2009 May;145(5):536-41. doi: 10.1016/j.surg.2009.01.012. PMID 19375613
- [Background] Huang MY, Scharf S, Chan PY. Effects of immersive virtual reality therapy on intravenous patient-controlled sedation during orthopaedic surgery under regional anesthesia: A randomized controlled trial. PLoS One. 2020 Feb 24;15(2):e0229320. doi: 10.1371/journal.pone.0229320. eCollection 2020. PMID 32092098
- [Background] Tolk JJ, Janssen RPA, Haanstra TM, van der Steen MMC, Bierma Zeinstra SMA, Reijman M. Outcome Expectations of Total Knee Arthroplasty Patients: The Influence of Demographic Factors, Pain, Personality Traits, Physical and Psychological Status. J Knee Surg. 2020 Oct;33(10):1034-1040. doi: 10.1055/s-0039-1692632. Epub 2019 Jul 4. PMID 31272124
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Kong H, West S. WMA DECLARATION OF HELSINKI - ETHICAL PRINCIPLES FOR Scienti c Requirements and Research Protocols. 2013; 29-32.
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. BMJ. 2007 Oct 20;335(7624):806-8. doi: 10.1136/bmj.39335.541782.AD. PMID 17947786
- [Background] Higgins JP, Altman DG, Gotzsche PC, Juni P, Moher D, Oxman AD, Savovic J, Schulz KF, Weeks L, Sterne JA; Cochrane Bias Methods Group; Cochrane Statistical Methods Group. The Cochrane Collaboration's tool for assessing risk of bias in randomised trials. BMJ. 2011 Oct 18;343:d5928. doi: 10.1136/bmj.d5928. PMID 22008217
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Shedden-Mora MC, Alberts J, Petrie KJ, Laferton JAC, von Blanckenburg P, Kohlmann S, Nestoriuc Y, Lowe B. The Treatment Expectation Questionnaire (TEX-Q): Validation of a generic multidimensional scale measuring patients' treatment expectations. PLoS One. 2023 Jan 23;18(1):e0280472. doi: 10.1371/journal.pone.0280472. eCollection 2023. PMID 36689398
- [Background] Sarah S, Lynn S. Is the Amsterdam Preoperative Anxiety and Information Scale (APAIS) a Valid Tool in Guiding the Management of Preoperative Anxiety in Adult Patients? A Literature Review. J Nurs Pract 2019; 3: 95-102.
- [Background] Baran O, Mordeniz C, Arar MC, Günkaya M. The Effect of Video Information on Preoperative Anxiety Levels in Patients Undergoing Total Knee Replacement. J Acad Res Med 2020; 10: 122-8.
- [Background] Celik F, Edipoglu IS. Evaluation of preoperative anxiety and fear of anesthesia using APAIS score. Eur J Med Res. 2018 Sep 11;23(1):41. doi: 10.1186/s40001-018-0339-4. PMID 30205837
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454